CLINICAL TRIAL: NCT02091817
Title: The Behavioral and Neural Effects of Oxytocin on Face Perception in Congenital Prosopagnosia
Brief Title: The Effect of Oxytocin on Face Perception
Status: Suspended | Phase: Early Phase 1 | Type: Interventional
Why Stopped: We are currently engaged in other behavioral study.
Sponsor: Soroka University Medical Center (Other)
Collaborators: Ben-Gurion University of the Negev (Other)
Responsible Party: Principal Investigator, Ilan Shelef, Head of medical imaging at Soroka University Medical Center, Soroka University Medical Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: sor010712ctil; ISF, 384/10 (Other Grant/Funding Number: israeli Science Foundation)
Record Dates: First submitted 2014-01-26; First posted 2014-03-19 (Estimated); Last update posted 2015-07-02 (Estimated); Status verified 2015-07

CONDITIONS: Healthy; Congenital Prosopagnosia
Keywords: oxytocin; face; memory
MeSH Terms: conditions — Prosopagnosia; Facies | interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (Other): Control group will be administered oxytocin and placebo, in a double-blind randomized order.
  Interventions: Drug: Oxytocin; Drug: Placebo
- congenital prosopagnosia (Experimental): Congenital prosopagnosics will be administered oxytocin and placebo in a double-blind randomized order.
  Interventions: Drug: Oxytocin; Drug: Placebo

INTERVENTIONS:
Drug: Oxytocin — Intervention will be examined on control group, and on experimental group as well.
  Other Names: syntocinon
Drug: Placebo — Placebo will be given to control group and experimental group as well.

SUMMARY:
The purpose of this study is to determine whether oxytocin affect face perception

ELIGIBILITY:
Inclusion Criteria:

* normal or corrected to normal vision

Exclusion Criteria:

* minors
* pregnancy (according to a pregnancy test taken by subjects prior to participation)
* a history of asthma or nasal polyps
* cardiac disorders
* hyponatremia
* acute or chronic renal insufficiency
* liver cirrhosis
* neurological disease
* other chronic disease
* dementia, or lack of judgment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2013-11; Primary Completion 2016-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Memory performance | Day 2 (24 hours after encoding)
  At the day participants will administer the substance, they will view a set of faces, of which they will be tested about 24 hours later. The measures that will be tested are %accuracy and %dwell time of eye movements towards each region in the faces the participants saw.

SECONDARY OUTCOMES:
Mood measurement | Day 1 (after oxytocin/placebo uptake)
  Participants will fill a PANAS mood questionnaire in order to monitor the effects of mood and fatigue of oxytocin/placebo. We will use ANOVA on the total score of the test in order to verify that differences in performance are not due to change in mood or fatigue after substance uptake.

CONTACTS AND LOCATIONS:
Overall Officials: Shelef Ilan, MD, Principal Investigator — Soroka University Medical Center; Galia Avidan, Ph.D, Principal Investigator — Ben-Gurion University of the Negev
Locations (1):
- Soroka medical center, Beersheba, Israel, Israel

REFERENCES:
- [Background] Avidan G, Behrmann M. Functional MRI reveals compromised neural integrity of the face processing network in congenital prosopagnosia. Curr Biol. 2009 Jul 14;19(13):1146-50. doi: 10.1016/j.cub.2009.04.060. Epub 2009 May 28. PMID 19481456
- [Background] Avidan G, Behrmann M. Implicit familiarity processing in congenital prosopagnosia. J Neuropsychol. 2008 Mar;2(1):141-64. doi: 10.1348/174866407x260180. PMID 19334309
- [Background] Avidan G, Hasson U, Malach R, Behrmann M. Detailed exploration of face-related processing in congenital prosopagnosia: 2. Functional neuroimaging findings. J Cogn Neurosci. 2005 Jul;17(7):1150-67. doi: 10.1162/0898929054475145. PMID 16102242
- [Background] Behrmann M, Avidan G, Marotta JJ, Kimchi R. Detailed exploration of face-related processing in congenital prosopagnosia: 1. Behavioral findings. J Cogn Neurosci. 2005 Jul;17(7):1130-49. doi: 10.1162/0898929054475154. PMID 16102241
- [Background] Hasson U, Avidan G, Deouell LY, Bentin S, Malach R. Face-selective activation in a congenital prosopagnosic subject. J Cogn Neurosci. 2003 Apr 1;15(3):419-31. doi: 10.1162/089892903321593135. PMID 12729493
- [Background] MacDonald E, Dadds MR, Brennan JL, Williams K, Levy F, Cauchi AJ. A review of safety, side-effects and subjective reactions to intranasal oxytocin in human research. Psychoneuroendocrinology. 2011 Sep;36(8):1114-26. doi: 10.1016/j.psyneuen.2011.02.015. Epub 2011 Mar 23. PMID 21429671
- [Background] Avidan G, Tanzer M, Hadj-Bouziane F, Liu N, Ungerleider LG, Behrmann M. Selective dissociation between core and extended regions of the face processing network in congenital prosopagnosia. Cereb Cortex. 2014 Jun;24(6):1565-78. doi: 10.1093/cercor/bht007. Epub 2013 Jan 31. PMID 23377287